CLINICAL TRIAL: NCT03549338
Title: A Ph2, Randomized, Open-Label, Multicenter, Three-Arm Trial of Sym004 Versus Each of Its Component Futuximab and Modotuximab, in Patients With Chemotherapy-Refractory Metastatic Colorectal Carcinoma and Acquired Resistance to Anti-EGFR mAb
Brief Title: Sym004 Versus Futuximab or Modotuximab in Patients With mCRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to administrative reasons
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-13; 2018-000618-39 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Cancer Metastatic; Carcinoma
Keywords: Metastatic Colorectal Cancer; Colorectal Cancer; Carcinoma; Sym004; futuximab; modotuximab
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma | interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Sym004) (Experimental): Sym004 will be given as a loading dose of 9 mg/kg on Cycle 1 Day 1 (C1D1), followed by weekly doses of 6 mg/kg beginning C1D8.
  For patients that crossover from Arm B and Arm C, Sym004 will be given at the dose level that contains the corresponding dose level of the respective individual antibody (futuximab or modotuximab) prior to crossover.
  Interventions: Drug: Sym004
- Arm B (Futuximab) (Experimental): Futuximab will be given as a loading dose of 4.5 mg/kg on C1D1, followed by weekly doses of 3 mg/kg beginning C1D8. At the End of Cycle 2 (EOC2), ongoing patients will crossover to Sym004; crossover may occur prior to the EOC2 in the event of early radiographic documentation of progressive disease (PD).
  Interventions: Drug: Futuximab
- Arm C (Modotuximab) (Experimental): Modotuximab will be given as a loading dose of 4.5 mg/kg on C1D1, followed by weekly doses of 3 mg/kg beginning C1D8. At the EOC2, ongoing patients will crossover to Sym004; crossover may occur prior to the EOC2 in the event of early radiographic documentation of PD.
  Interventions: Drug: Modotuximab

INTERVENTIONS:
Drug: Sym004 — Sym004 is a 1:1 mixture of two recombinant mAbs (futuximab and modotuximab) which bind specifically to non-overlapping epitopes located in the extracellular domain (ECD) of the EGFR.
  Arms: Arm A (Sym004)
Drug: Futuximab — Futuximab is one of two mAb components that constitute Sym004.
  Arms: Arm B (Futuximab)
Drug: Modotuximab — Modotuximab is one of two mAb components that constitute Sym004.
  Arms: Arm C (Modotuximab)

SUMMARY:
This is a Phase 2, randomized, open-label, 3-arm trial in the ratio of 1:1:1 to either Sym004 (Arm A) versus each of its component monoclonal antibodies (mAbs), futuximab (Arm B) or modotuximab (Arm C), in genomically-selected patients with chemotherapy-refractory metastatic colorectal carcinoma (mCRC) and acquired resistance to anti-epidermal growth factor receptor (anti-EGFR) mAb therapy. The study is designed to evaluate the relative antitumor activity of each agent as assessed by imaging studies performed after 8 weeks of treatment.

DETAILED DESCRIPTION:
Following consent and prior to randomization, genomic analysis will be conducted on blood samples obtained from each potential patient. Triple-negative (TN) results as defined in trial eligibility criteria will be required for initial eligibility. Patients with TNmCRC will continue in the screening process. Once deemed fully eligible, patients will be randomized to Arm A, Arm B, or Arm C.

Dosing cycles of 28 days will continue until documented disease progression (PD) or another criterion for discontinuation is met. Antitumor activity will be assessed at the end of every 2 cycles (every 8 weeks [Q8W]). At the End of Cycle 2 (EOC2) tumor assessment:

* Patients assigned to Arm A (Sym004) with a documented objective response (OR) or stable disease (SD) will continue to receive Sym004; patients at the EOC2 with documented PD will be discontinued from study
* Patients assigned to Arm B (futuximab) or Arm C (modotuximab) with a documented OR or SD will be crossed-over to receive Sym004; patients with documented PD at the EOC2 (or prior to the EOC2) will be offered the opportunity to crossover to receive Sym004 or will be discontinued from study

To be considered evaluable for antitumor activity assessment, patients must have completed 2 cycles of dosing inclusive of EOC2 disease imaging studies and must have received any amount of their assigned investigational medicinal product (IMP) during that period, or have PD documented by imaging studies prior to the EOC2. Non-evaluable patients and patients discontinuing from study prior to the EOC2 for reasons other than documented PD will not be replaced.

Note: In December 2018, the decision was made to terminate the trial and enrollment was prematurely discontinued. The primary, secondary, and exploratory objectives are no longer applicable. Only clinical safety-related evaluations will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age at the time of obtaining informed consent.
* Histologically- or cytologically-confirmed mCRC.
* Microsatellite instability-high (MSI-H) / mismatch repair-deficient (dMMR) tumors must have received prior therapy with pembrolizumab, nivolumab, or other programmed cell death protein-1 (PD-1)/programmed death-ligand 1 (PD-L1) pathway blocker, and must have progressed on that therapy.
* Meeting the protocol definition of TNmCRC assessed in the screening blood test.
* mCRC currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
* Measurable disease according to RECIST v1.1, and willingness to undergo a total of 2 biopsies of a primary or metastatic tumor site(s) considered safely accessible for biopsy.
* Must have received at least 2 prior regimens of standard chemotherapy for mCRC and must have been refractory to or failed (includes intolerance to) those regimens. Prior standard chemotherapy may not have included TAS-102 or regorafenib, but must have included agents as specified in the protocol.
* "Acquired" resistance to commercially available anti-EGFR mAbs approved for the treatment of mCRC must have:

  1. Received treatment with an anti-EGFR for ≥16 weeks
  2. Progressive disease (PD) documented by imaging or clinical findings less than or equal to 6 calendar months after cessation of previous anti-EGFR mAb treatment
  3. No more than 6 calendar months from last dose of previous anti-EGFR mAb treatment to date of consent for this trial (regardless of the line of therapy in which it was used)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Not of childbearing potential or who agree to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 3 months after the last dose of study drug.

Exclusion Criteria:

* Women who are pregnant or lactating or intending to become pregnant before, during, or within 3 months after the last dose of study drug.
* Prior history of specific mutations (specified in the protocol) in the tumor at the time of any previous assessment.
* Known, untreated central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression; patients with any of these not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required
* An active second malignancy or history of another malignancy within the last 5 years, with exceptions.
* Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to first administration of study drug unless adequately treated and considered by the Investigator to be stable.
* Active uncontrolled bleeding or a known bleeding diathesis
* Known clinically significant cardiovascular disease or condition.
* Non-healing wounds on any part of the body.
* Significant gastrointestinal abnormality.
* Skin rash > Grade 1 from prior anti-EGFR therapy at the time of randomization.
* Unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy

Drugs and Other Treatments Exclusion Criteria:

* Prior treatment with TAS-102 or regorafenib
* Any antineoplastic agent for the primary malignancy (standard or investigational) without delayed toxicity within 4 weeks prior to first administration of IMP and during study with exceptions
* Any other investigational treatments within 4 weeks prior to and during study; includes participation in any medical device or other therapeutic intervention clinical trials
* Radiotherapy as specified in the protocol
* Immunosuppressive or systemic hormonal therapy (> 10 mg daily prednisone equivalent) within 2 weeks prior to first administration of IMP and during study; allowed therapies are specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD,PhD,FACP, Principal Investigator — M.D. Anderson Cancer Center
Locations (18):
- United States (5):
  - City of Hope - Comprehensive Cancer Center, Duarte, California
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (5):
  - Uniklinik Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Asklepios Kliniken Altona, Hamburg
  - Universitätsmedizin Mannheim, Mannheim
  - Städtisches Klinikum München, München
- Italy (3):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Università degli Studi della Campania "Luigi Vanvitelli", Napoli
- Spain (5):
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intended number of patients to be included in this trial was approximately 54 (18 evaluable per Arm). As of the trial termination date, 2 patients were enrolled.
Pre-assignment Details: The first patient was randomized to Arm B prior to the trial termination date and crossed over to Sym004 at the EOC1. The second patient was randomized to Arm B after the trial termination date, but enrolled to Arm A per Sponsor decision.
Period: Overall Study
Arm/Group | Arm A (Sym004) | Arm B (Futuximab) | Arm C (Modotuximab)
Started | 1 | 1 | 0
Completed | 0 | 0 (Patient crossed-over to Sym004 at the EOC1 per Sponsor decision following trial termination.) | 0
Not Completed | 1 | 1 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Clinical Progression | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients were treated in Arm C due to the early termination of the trial.
Groups:
- Arm A (Sym004): Sym004 will be given as a loading dose of 9 mg/kg on Cycle 1/Day 1 (C1D1), followed by weekly doses of 6 mg/kg beginning C1D8.
- Arm B (Futuximab): Futuximab will be given as a loading dose of 4.5 mg/kg on C1D1, followed by weekly doses of 3 mg/kg beginning C1D8. At the End of Cycle 2 (EOC2), ongoing patients will be crossed-over to Sym004; crossover may occur prior to the EOC2 in the event of early radiographic documentation of progressive disease (PD). Sym004 will be given at the dose level that contains the corresponding dose level of the individual antibody futuximab prior to crossover.
- Arm C (Modotuximab): Modotuximab will be given as a loading dose of 4.5 mg/kg on C1D1, followed by weekly doses of 3 mg/kg beginning C1D8. At the EOC2, ongoing patients will be crossed-over to Sym004; crossover may occur prior to the EOC2 in the event of early radiographic documentation of PD. Sym004 will be given at the dose level that contains the corresponding dose level of the individual antibody modotuximab prior to crossover.
- Total: Total of all reporting groups
Arm/Group | Arm A (Sym004) | Arm B (Futuximab) | Arm C (Modotuximab) | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 1 | 1 |  | 2
  >=65 years | 0 | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 |  | 0
  Male | 1 | 1 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 1 | 1 |  | 2
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 1 | 1 |  | 2
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) by Nature, Severity, and Occurrence.
Description: Measured From Baseline to End of Trial Participation, as Assessed by the Common Terminology Criteria for AEs (Version 5) (CTCAE v5). AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) terminology and the severity of the toxicities will be graded according to the CTCAE v5, where applicable.
Time Frame: 4 months
Population: The first patient was randomized to Arm B prior to the trial termination date and crossed over to Sym004 at the EOC1. The second patient was randomized to Arm B after the trial termination date, but enrolled to Arm A per Sponsor decision.
Measure: Number; unit: participants
Arm/Group | Arm A (Sym004) | Arm B (Futuximab)
Number analyzed (Participants) | 2 | 1
participants
  At least one AE | 2 | 1
  At least one SAE | 1 | 0
  At least one AE related to Sym004 | 2 | 0
  At least one AE related to futuximab | 0 | 0
  At least one SAE related to Sym004 | 0 | 0
  At least one SAE related to futuximab | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Arm A (Sym004) | Arm B (Futuximab)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sym004) (N=2) | Arm B (Futuximab) (N=1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sym004) (N=2) | Arm B (Futuximab) (N=1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination changed the primary objective to assess the safety of the allocated treatment. Collection of data for secondary and exploratory objectives was omitted. The crossover dose plan as detailed was no longer in effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication before the completion of the trial without written approval from the Sponsor. Publications shall not disclose any Sponsor confidential information and property (not including the trial results). The Sponsor reserves the right to review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT03549338/Prot_000.pdf